CLINICAL TRIAL: NCT02629484
Title: A Pilot Study to Assess Feasibility, Compliance, Safety and Group Separation for a Multicentre Randomised Trial of Preoperative Focused Cardiac Ultrasound for Fractured Neck of Femur Surgery
Brief Title: Trial of Focused Cardiac Ultrasound for Fractured Neck of Femur Surgery
Acronym: ECHONOFII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Melbourne (Other)
Collaborators: Melbourne Health (Other); Austin Health (Other Government)
Responsible Party: Principal Investigator, Colin Royse, Professor of Anaesthesia, University of Melbourne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2015.231
Record Dates: First submitted 2015-12-01; First posted 2015-12-14 (Estimated); Last update posted 2018-05-02 (Actual); Status verified 2018-04

CONDITIONS: Hip Fractures
Keywords: echocardiography; hip fracture; surgery; outcomes
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Focused Cardiac Ultrasound (Active Comparator): participants randomised to receive focused cardiac ultrasound prior to surgery for hip fracture
  Interventions: Other: Focused cardiac ultrasound
- Standard care (clinical assessment) (No Intervention): Participants randomised to standard care receive clinical assessment of the patient

INTERVENTIONS:
Other: Focused cardiac ultrasound — focused cardiac ultrasound is a goal-focused transthoracic echocardiography examination of the heart, aimed to improve the diagnostic accuracy of clinical assessment
  Arms: Focused Cardiac Ultrasound

SUMMARY:
Hip fracture surgery is a major world health care burden and concern, as it has a large and increasing prevalence and carries very high patient mortality, disability and community health care cost. As the commonest cause of mortality is from cardiac complications, and cardiac disease is prevalent and frequently missed by standard care, we hypothesise that earlier and more accurate diagnosis and treatment of cardiac pathology in this cohort will lead to improved outcome. Focused cardiac ultrasound (FCU) is a new increasingly popular technique used by doctors that enables earlier and more accurate diagnosis of cardiac disorders that can be performed routinely before hip fracture surgery. Our preliminary data of 64 patients demonstrated that routine FCU before surgery lead to a change in cardiac diagnosis and management in 50% of patients requiring hip fracture surgery, which was associated with a 50% reduction in mortality 12 months after surgery compared with controls. It is therefore important for a large randomised trial to be performed to confirm or rebuke these findings, as if true, would have a very large impact on health care and may also improve health care and outcome in other high-risk surgical populations. The proposed pilot study is a pilot study which aims to establish feasibility, safety, compliance and group separation prior to commencing a definitive multicentre trial.

DETAILED DESCRIPTION:
Aims and Hypotheses Aims

1. To determine whether routine preoperative focused cardiac ultrasound (FCU) leads to a reduced composite outcome of death, major adverse cardiac events, and acute renal failure (adverse composite outcome) 30 days after hip fracture surgery compared to patients who do not receive preoperative FCU (current standard of care).
2. To identify the changes in team management of the patient due to FCU that are associated with improved outcome, compared to current standard of care.
3. To determine whether routine preoperative FCU is more cost-effective than current standard of care.

Hypotheses

1. FCU reduces adverse composite outcome by at least 20%, 30 days after hip fracture surgery.
2. FCU leads to changes in cardiac diagnosis, and subsequent changes to perioperative and post-discharge management plans, which are associated with improved outcome compared to current standard of care.
3. Routine FCU before hip fracture surgery is more cost-effective than current standard of care.

Identifying cardiovascular disease: Preoperative cardiac assessment, which enables improved cardiac treatment and reduction of cardiac complications, is recommended by the American Heart Association. However, cardiovascular disease is often unrecognised and under-diagnosed in this age group because of frailty, general immobility, and the high frequency of poor cognitive function including dementia, which inhibits accurate clinical assessment. Careful cardiac assessment and treatment is often not undertaken because of the belief that surgery should be performed urgently and a delay for cardiac investigations may worsen outcome.

Cardiac risk factors for death after hip fracture surgery (cardiac failure, aortic stenosis, pulmonary hypertension and right ventricular hypertrophy) cannot be reliably diagnosed with clinical examination and require echocardiography (FCU or transthoracic echocardiography (TTE)). Although a pulmonary embolus cannot be reliably diagnosed with echocardiography, the haemodynamic effects from a significant pulmonary embolus are readily seen (right ventricular dilatation and failure). Currently, preoperative TTE is only used in selected patients, based on the clinical assessment and the opinion of the clinician as to whether it is justified. If the anaesthetist reviews the patient just prior to surgery and is concerned about cardiovascular disease, there is a lot of pressure to proceed with booked surgery due to the current belief that early surgery saves lives, rather than to delay surgery for a TTE. Treatment is therefore often based on "best guess" clinical assessment. This management approach may lead to inadequate treatment with resultant hypotension, leading to organ failure and death.

Focused Cardiac Ultrasound (FCU): The conventional TTE investigation is ordered by the treating doctor, performed by a technician and reported by a cardiologist or radiologist at a later time. The TTE provides detailed information on structure and function of all of the valves and chambers and is also referred to as diagnostic echocardiography. A TTE or other complex cardiovascular investigation leads to delay, as the process of obtaining a TTE and then waiting for the report may take days depending on resource availability. Any echocardiography examination is a "snapshot" in time, and heart function can change between the performance of the TTE and the commencement of surgery. A FCU utilises the same echocardiography techniques as conventional TTE but is performed as a bedside test by the treating doctor to answer a clinical question to aid clinical decision-making in real time. It provides specific information relevant to perioperative care in time for acute resuscitation and potentially life-saving decision-making.

A type of FCU, iHeartScanTM , that is specifically designed for critical and perioperative care has been developed by the Ultrasound Education Group at The University of Melbourne. FCU has been confirmed to be as accurate as comprehensive TTE for purposes of acute clinical care. FCU has been endorsed by The American Society of Echocardiography and embraced by the critical care community.

The case for equipoise: The conventional approach to proceed to early surgery without delay for cardiovascular investigations is contrary to the proof-of-concept data that preoperative FCU may reduce mortality through the provision of better cardiovascular diagnostic information, leading to management changes. The use of conventional TTE, however, causes considerable delay to surgery, which may increase mortality risk. FCU has the advantage of providing improved diagnosis without causing substantial delay to surgery, and can therefore is additive to rather than competitive with current "best practice". An economic analysis of routine FCU has not been performed.

Feasibility of the trial - the ECHONOF II trial In the preliminary study, feasibility of routine FCU in hip fracture surgery was demonstrated, with more than one patient per week at one centre. To determine feasibility of the proposed outcome randomised controlled trial (RCT) a pilot study of feasibility, safety, protocol compliance and group separation will be conducted in 2016 at 4-5 sites across Australia, with the lead site at Royal Melbourne Hospital. The pilot study analysis will include patients recruited who have 30-day data available a in 2016, though data will continue to be collected out to 12 months.

The pilot study protocol will be the same as the proposed (future) definitive clinical trial , but the endpoints are aimed at assessing feasibility and compliance.

1. Feasibility outcomes

   1. the number of patients screened: recruited ratio < 4:1
   2. recruitment rate of 1 patient/week/centre
2. Safety

   1. No harm to patients from performing FCU
   2. No surgical delay > 1 hour by waiting for FCU to be performed
3. Protocol Compliance

   1. FCU performed < 24 hrs. of surgery
   2. Treating team notified of FCU result
   3. Follow up at all time points (unless death)
   4. Incidence of comprehensive TTE in standard group before and after surgery
   5. Adverse complications adjudication performed by the adjudication committee
4. Group separation

   1. Completion of preoperative and actual perioperative management plans in both groups
   2. Analysis for difference in diagnosis and management between groups: aim > 20% difference between groups

Research protocol Trial Design: A parallel group, randomised controlled, multicentre trial with 1:1 allocation ratio.

Participants: Patients presenting with isolated, primary, non-metastatic fractured neck of femur, where surgery is expected within 48 hours after hospital admission will be recruited. Patients with prior hip surgery on the affected side, or where the cause is likely to be due to metastatic cancer, or where survival is unlikely in the 24 hours from admission will not be included.

Settings and Locations: teaching and regional hospitals in Australia with a high volume of hip fracture surgery and the necessary equipment and expertise to perform FCU have agreed to participate.

Intervention: Participants randomised to the FCU group will receive a preoperative FCU performed by an independent operator within 24 hours of planned surgery, following The University of Melbourne iHeartScanTM protocol. Patients randomised to the standard care group will not undergo FCU before surgery.

There are no restrictions on the treating team in either group determining what management they will employ, including anaesthesia technique, surgical management, perioperative care and preoperative investigations including comprehensive TTE by the cardiology department. However the treatment of patients will be recorded, allowing comparison of the effect of FCU on diagnosis and management between groups.

The control group will represent the standard of care in each of the participating hospitals. This typically includes early surgery with minimal preoperative investigations. Some patients, however, based on the clinical assessment of their treating doctors, will have additional investigations such as comprehensive TTE, which could result in changes in management including an associated delay in surgery. This trial will not interfere with the standard of care management, and, once recruited, patients will remain in the standard of care group even if they receive comprehensive TTE or have delayed surgery. Treatment in both groups will be according to individual and institutional practice, working with the diagnostic information available at the time.

Randomisation: Randomisation codes will be in blocks using a web-based automatic enrolment system to participating institutions in order to facilitate recruitment across different time zones and out-of-hours cases. Patients will be stratified to severity of surgery (hip replacement/hemiarthroplasty, or femoral fixation) and institution (tertiary referral, or non-tertiary metropolitan/ regional hospitals). The randomisation sequence will be generated using a computer random sequence generator for each strata in blocks of 10 to ensure close balance of the numbers in each group at any one time during the trial.

Allocation concealment and implementation: The allocation sequence will be concealed by the web-based enrolment system. The site research staff will recruit patients and organise an in dependent practitioner to perform FCU (or not). The independent practitioner will receive the allocation and whether to perform FCU or not, and place the completed or blank FCU form in a sealed envelope. The treating doctors will first complete a management plan before opening the envelope to obtain the completed or blank FCU form. The FCU form will then be placed in a second sealed envelope which is not opened until the allocation sequence is revealed. The research staff who will collect outcome data are not involved in patient recruitment and will therefore be blinded to group allocation. The central trial monitor who adjudicates outcomes with the assistance of 2 clinicians are also blinded to allocation.

Statistical methods: The Statistical Consulting Group (University of Melbourne), supervised by team statistician Dr Sandy Clarke,will advise and supervise statistical methods, data management, integrity, security and analysis. The primary outcome will be compared between FCU and control groups using binary logistic regression, with the control group as the reference category. The survival times will be analysed using Cox proportional hazards regression. A pre-determined sub-group analysis will separate those with and without an existing TTE in the previous 12 months. Relative risk of death will be analysed using Cox proportional hazard regression. Patterns of management and relative risk (of death) will be compared between groups using a two-sample t-test including sub-group analysis of pathology identified by FCU (e.g., hypovolaemia, cardiac failure and aortic stenosis).

Clinical trial coordination: The trial will be managed through the Department of Surgery, The University of Melbourne. This will include all aspects of trial control, data collation, and site co-ordination. An independent committee including a statistician, clinical trial monitor, clinician, and member of the Melbourne Health Human Research Ethics Committee will oversee trial safety and data integrity. The committee will perform a planned, blinded interim analysis, after 50% recruitment.

Endpoint adjudication committee An end point committee consisting of a trial monitor and 2 clinicians, blinded to treatment allocation, will be established to adjudicate the non-fatal cardiovascular events at 6 monthly intervals. This committee will also advise on event rate, (blinded) group separation, feasibility and stopping rules.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with isolated, primary, non-metastatic fractured neck of femur, where surgery is expected within 48 hours after hospital admission will be recruited.

Exclusion Criteria:

* Patients with prior hip surgery on the affected side, or where the cause is likely to be due to metastatic cancer, or where survival is unlikely in the 24 hours from admission will not be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2017-01-26 (Actual); Study Completion 2018-01-26 (Actual)

PRIMARY OUTCOMES:
Composite mortality and morbidity score | 30 days after surgery
  The primary outcome is 30 day composite outcome of the incidence of mortality, acute kidney injury, and cardiovascular morbidity (including non-fatal myocardial infarction, stroke, pulmonary embolism or cardiac arrest.

SECONDARY OUTCOMES:
The number of days alive, out of hospital, and until return to place of origin | 12 months
  Longitudinal measures include the number of days alive, out of hospital and returning to their place of origin out to 12 months.
Changes in clinician diagnosis and management from a recorded preoperative plan | 30 days
  The treating doctors will complete a diagnosis and management research form prior to revealing the FCU findings or not. The actual management of the patient after allocation will be recorded prospectively for all patients, with the data recording sheets not showing allocation. Data include cardiac monitoring and treatment preoperatively, intraoperatively and postoperatively, including type of anaesthesia, fluid therapy, inotropes, other invasive organ support and intensive care use, surgical technique, and additional cardiovascular management post-hospital discharge.
Total cost of care | 12 months
  Units of health care resources consumed will be combined with Australian unit costs derived from Pharmaceutical benefit schedule, Medicare and Australian Diagnostic group indicators. The dollar value for each component of stay (e.g. days in hospital, drugs used, investigations performed) will be converted into a cost value and aggregated to make a single cost over the 12 month follow up period
EuroQol Health status score | 12 months
  The EuroQol health status survey instrument is a a standard, internationally validated instrument with Australian population norms, will be conducted at 12 months follow up

CONTACTS AND LOCATIONS:
Overall Officials: Colin Royse, MD, BS, Principal Investigator — University of Melbourne
Locations (3):
- Australia (3):
  - Prince Charles Hospital, Brisbane, Queensland
  - Royal Melbourne Hospital, Melbourne, Victoria
  - Western and Sunshine General hospitals, Melbourne, Victoria